CLINICAL TRIAL: NCT06027216
Title: Monocular Visual Confusion for Field Expansion
Brief Title: Multiplexing Prism Fitting for Field Expansion of Monocular Vision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Eli Peli, Senior Scientist, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2023P001878; R01EY031777 (NIH)
Record Dates: First submitted 2023-08-29; First posted 2023-09-07 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: One Eye Blindness; Blind Left Eye; Blind Right Eye
Keywords: Field expansion; Collision detection; Walking; Response time
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Intervention Model Description: Individuals with Acquired Monocular Vision/ Blindness in One Eye
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Field Expansion (Experimental): Field of view on the nasal side (same side as the blind eye) with and without multiplexing prism
  Interventions: Device: Multiplexing Prism

INTERVENTIONS:
Device: Multiplexing Prism — Multiplexing prism is designed for spatial vision multiplexing. It allows partial light transmission through the prism allow the observer to simultaneously see the physical world through the prism and see the "shifted view" from the non-seeing side. It is developed to expand the field of view of individuals with just one eye.

SUMMARY:
The investigators are developing an assistive device, known as multiplexing prism that expands the field of view for individuals with acquired monocular vision (loss of an eye). The investigators are testing a simplified design and fitting protocol to provide field expansion for individuals with acquired monocular vision.

ELIGIBILITY:
Inclusion Criteria:

* No medical health issues such as seizures, motor movements problem
* Loss of vision in one eye (less than 20/200) for >1 year)
* Visual acuity of the seeing eye: Better than 20/32 visual acuity with correction
* No visual field defect in the seeing eye (nasal field of at least >45degree)
* No medical health issues such as seizures, motor movements problem

Exclusion Criteria:

* Patients with any physical or mental disabilities, including cognitive dysfunction, balance problems, or other deficits that could impair their ability to respond to the stimuli presented in this study will be excluded
* Any person with motor movements problem (e.g., unable to use extremities)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eli Peli, OD, Principal Investigator — Schepens Eye Research Institute
Locations (1):
- Schepens Eye Research Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jung JH, Peli E. Field Expansion for Acquired Monocular Vision Using a Multiplexing Prism. Optom Vis Sci. 2018 Sep;95(9):814-828. doi: 10.1097/OPX.0000000000001277. PMID 30169357
- [Background] Jung JH, Peli E. No Useful Field Expansion with Full-field Prisms. Optom Vis Sci. 2018 Sep;95(9):805-813. doi: 10.1097/OPX.0000000000001271. PMID 30169356
- [Background] Peli E, Jung JH. Multiplexing Prisms for Field Expansion. Optom Vis Sci. 2017 Aug;94(8):817-829. doi: 10.1097/OPX.0000000000001102. PMID 28727615

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled Participants for Multiplexing Prism: Of the 30 enrolled participants, 22 met the inclusion criteria and were prescribed with the multiplexing prism.
Period: Overall Study
Arm/Group | Enrolled Participants for Multiplexing Prism
Started | 30
Completed | 22
Not Completed | 8
Not completed — Did not qualify | 8

BASELINE CHARACTERISTICS:
Groups:
- Patient's Demography: Adult individual with acquired monocular vision (seeing with one eye)
Arm/Group | Patient's Demography
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Nasal Visual Field of the Seeing/Functioning Eye [Mean (Standard Deviation); unit: degree] | 55 (4)

OUTCOME MEASURES:

1. Primary Outcome: Gain in Visual Field With the Multiplexing Prism
Description: Field expansion is calculated based on the difference of the maximum field of view on the nasal side of the seeing/functioning eye (same side as the blind eye) with and without multiplexing prism.
Time Frame: Visit 2 of Study (approximately 2-3 weeks after 1st Visit)
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Amount of Visual Field Expansion: The maximum field of view on the nasal side (same side as the blind eye) of the participants with and without the multiplexing prism is measured. An increase in visual field indicates field expansion/gain.
Arm/Group | Amount of Visual Field Expansion
Number analyzed (Participants) | 22
degrees | 24 (4)

2. Secondary Outcome: Maximum Extent of Nasal Visual Field With the Multiplexing Prism
Description: The farthest extent of the nasal visual field with the multiplexing prism placed in front of the seeing eye.
Time Frame: Visit 2 of Study (approximately 2-3 weeks after 1st Visit)
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Nasal Visual Field With the Multiplexing Prism: The baseline nasal field of the seeing eye is 55 degrees (±4) without the multiplexing prism.
Arm/Group | Nasal Visual Field With the Multiplexing Prism
Number analyzed (Participants) | 22
degrees | 79 (5)

ADVERSE EVENTS:
Time Frame: The end of Visit 1 and Visit 2.
Description: The intervention only involves a magnetic clip-on multiplexing prism that can be attached/removed easily from a pair of glasses, with minimal risks.
Groups:
- Patient's Demography: Adult individuals with acquired monocular vision (seeing with one eye)
Arm/Group | Patient's Demography
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT06027216/Prot_SAP_000.pdf